CLINICAL TRIAL: NCT02115750
Title: A Double-Blind, Randomized, Parallel-Group, Active-Control Study to Compare the Efficacy and Safety of CHS-0214 Versus Enbrel in Subjects With Rheumatoid Arthritis and Inadequate Response to Treatment With Methotrexate
Brief Title: Comparison of CHS-0214 to Enbrel (Etanercept) in Patients With Rheumatoid Arthritis (RA)
Acronym: CHS-0214-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS-0214-02
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis
Keywords: CHS-0214; Enbrel; RA; Biosimilar; Etanercept
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enbrel (etanercept) (Active Comparator): Enbrel 50mg weekly times 24 weeks.
  Interventions: Drug: Etanercept
- CHS-0214 (Experimental): CHS-0214 50mg weekly times 24 weeks.
  Interventions: Drug: CHS-0214

INTERVENTIONS:
Drug: Etanercept — Head-to-head comparison
  Other Names: Enbrel; European Enbrel
  Arms: Enbrel (etanercept)
Drug: CHS-0214
  Arms: CHS-0214

SUMMARY:
This is a two part study comparing CHS-0214 to Enbrel in patients with active rheumatoid arthritis and an inadequate response with Methotrexate (MTX) who are naive to biologic therapies.

Pt.1 is a 24-week randomized, double-blind, active-control, parallel-group, multi-center global study. The primary end point is 20% improvement in American College of Rheumatology criteria (ACR-20) at week 24. Comparing CHS-0214 to Enbrel for efficacy and safety.

Pt. 2 is an open-label single arm study in which patients with at least an ACR-20 response receive CHS-0214. Continued response and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults
* RA (Rheumatoid Arthritis) diagnosis for 6 months
* On stable dose of MTX of 8mg to 25mg per week
* Active disease: greater than 6 tender joints, greater than 6 swollen joints, C-reactive protein (CRP) greater than or equal to 0.5mg/dL, and disease activity score (DAS) with 28 joints (DAS28-CRP(4)) greater than or equal to 3.2

Exclusion Criteria:

* Use of prednisone greater than 10mg/day
* Use of greater than one non-steroidal anti-inflammatory drug (NSAID)
* Use of biologic therapies for any cause
* Chemistry and hematology values outside protocol specified range
* Positive QuantiFERON-tuberculosis (TB) Gold Test
* Evidence of active lung disease on chest x-ray
* Major systemic infections
* Presence of significant comorbid conditions
* Known allergy to latex
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Finck, M.D., Study Director — Coherus Oncology, Inc.
Locations (141):
- United States (37):
  - Elite Clinical Studies, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Dream Team Clinical Research, Anaheim, California
  - Advanced Medical Research, Lakewood, California
  - Pro Health Partners, Long Beach, California
  - St. Joseph Hospital of Orange, Orange, California
  - Desert Medical Advances, Palm Desert, California
  - Kaiser Permanente - CA, Richmond, California
  - Med Investigators, Inc, Roseville, California
  - Troum Medical Associates, Santa Monica, California
  - Inland Rheumatology Clinical Trials Inc, Upland, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Hope Clinical Research, Kissimmee, Florida
  - Advanced Medical Research, Inc, Orlando, Florida
  - Allergy & Rheumatology Associates LLC, St. Petersburg, Florida
  - HealthPoint Medical Group, Tampa, Florida
  - Bluegrass Community Research, Inc, Lexington, Kentucky
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Arthritis Center of Nebraska, Lincoln, Nebraska
  - Pacific Arthritis Center Medical Group, Omaha, Nebraska
  - Rheumatoid Arthritis Investigational Network, Omaha, Nebraska
  - North Shore University Hospital, Great Neck, New York
  - Montefiore Medical Center, The Bronx, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - PMG Research of Wilmington LLC, Wilmington, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Low Country Rheumatology, Charleston, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - Texas Physicians Medical Research Group, Arlington, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Pioneer Research Solutions Inc, Houston, Texas
  - Arthritis Northwest Rheumatology PLLC, Spokane, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin
  - Gundersen Lutheran Medical Center, Onalaska, Wisconsin
- Belarus (6):
  - Brest Regional Clinical Hospital, Brest
  - Grodno Regional Clinical Hospital, Grodno
  - Gomel Regional Clinical Hospital, Homyel
  - City Clinical Hospital #1 - Belarus, Minsk
  - City Clinical Hospital #9 - Belarus, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- France (5):
  - Hôpital Michallon - CHU de Grenobl, Grenoble
  - CHU Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional D'Orleans, Orléans
  - Hopital Cochin-Saint Vincent de Paul, Paris
  - Hopital de Saint Etienne, Saint-Etienne
- Germany (5):
  - Asklepios Klinikum Bad Abbach, Bad Abbach
  - Klinische Forschung Dresden GmbH, Dresden
  - Center of Innovative Diagnostics and Therapeutics Rheumatology/Immunology, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - SMO.MD GmbH - Zentrum fuer klinische Studien, Magdeburg
- Hungary (7):
  - St. Rokus Hospital, BAJA, Baja
  - DRC Gyogzszervizsgalo Kozpont, Balatonfüred
  - Orszagos Reumatologiai es Fizioterapias Intezet, Budapest
  - Qualiclinic Kft, Budapest
  - Békés Megyei Pándy Kálmán Kórház, Gyula
  - University of Szeged, Faculty of Medicine, Szeged
  - Rakoczi Ferenc Korhaz-CRU Hungary (KFT), Szikszó
- Israel (4):
  - Rambam Medical Center, Haifa
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Ẕerifin
- Japan (40):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Inoue Hospital, Takasaki-shi, Gunma
  - Hiroshima Clinic, Nishiku, Hiroshimashi
  - Izumi Himawari Clinica, Sendai, Miyagi
  - Miyashita Rheumatology Clinic, Omura-shi, Nagasaki
  - Japanese Red Cross Okayama Hospital, Okayama, Okayama-ken
  - Japanese Red Cross Nagoya Daiichi Hospital, Aichi
  - Yamada Rheumatology Clinic, Ehime
  - University of Occupational and Environmental Health Hospital, Fukuoka
  - Kondo Clinic for Rheumatism and Orthopaedics, Fukuoka
  - Medical Co. LTA PS Clinic, Fukuoka
  - Shono Rheumatism Clinic, Fukuoka
  - St Mary;s Hospital, Fukuoka
  - Hiroshima Rheumatology Clinic, Hiroshima
  - Medical Corporation Nakayama Clinic, Hyōgo
  - Matsubara Mayflower Hospital, Hyōgo
  - Eiraku Clinic, Kagoshima
  - Izumihara Rheumatic and Medical Clinic, Kagoshima
  - Kawasaki Rheumatism and Internal Medicine Clinic, Kanagawa
  - Kumamoto Orthopaedic Hospital, Kumamoto
  - Munakata Yasuhiko Clinic, Miyagi
  - Yu-Family Clinic, Miyagi
  - Sendai Taihaku Hospital, Miyagi
  - Kai Clinic, Miyazaki
  - Zenjinkai Shimin no Mori Hospital, Miyazaki
  - Komagamine Orthopaedic Rheumatic Clinic, Morioka Iwate
  - Nagasaki Medical Hospital of Rheumatology, Nagasaki
  - Nagasaki University Hospital, Nagasaki
  - SaSebo Chuo Hospital, Nagasaki
  - Yoshida Orthopaedic and Rheumatology Clinic, Numakunai
  - Rinku Hashimoto Rheumatology Orthopedics, Osaka
  - Oribe Clinic of Rheumatism and Medicine, Ōita
  - Otsuka Clinica of Rheumatism and Medicine, Ōita
  - Koshigaya Municipal Hospital, Saitama
  - Medical Corporation Kojyokai Hirose Clinic, Saitama
  - Hokkaido Medical Center for Rheumatic Diseases, Sapporo
  - St. Luke's International Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Miyasato Clinic, Yamaguchi
  - Tokito Clinic Rheumatology and Orthopaedics, Surgery, Yamaguchi
- Poland (13):
  - Centrum Kliniczno Badawcze, Elblag
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Mazowieckie Centrum Badan Klinicznych (MCBK) SC, Grodzisk Mazowiecki
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Centrum Terapii Wspólczesne, Kodz
  - NZOZ Lecznica MAK-MED, Nadarzyn
  - Profmedicus sp. z o.o, Olsztyn
  - Centrum Medyczne SYNEXUS Poznan, Poznan
  - Prywatna Praktyka Lekarska Prof UM dr hab. Med. Pawel Hrycaj, Poznan
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - Biogenes NZOZ, Wroclaw
  - Synexus Polska Sp. z o.o, Wroclaw
- Russia (10):
  - Krasnoyarsk Medical Academy, Krasnoyarsk
  - State Healthcare Institution of Moscow City Clinical Hospital #15 n.a. O.M. Filatov, Moscow
  - Practicheskaya Meditsina, Ltd, Moscow
  - Republican Hospital n.a. V.A. Baranov, Petrozavodsk
  - Medical Research Institute, LLC, Saint Petersburg
  - St. Petersburg State Healthcare Institution "Consultative diagnostic center #85, Saint Petersburg
  - Smolensk State Medical University (SSMU), Smolensk
  - Municipal Healthcare Institution "Emergency Clinical Hospital n.a. N.V. Soloviev, Yaroslavl
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
  - MBI "Central City Clinical Hospital #6, Yekaterinburg
- South Africa (8):
  - Dr CI Louw, Cape Town
  - Dr S Nayiager, Durban
  - Wits Donald Gordon Clinical Trial Site, Johannesburg
  - Drs Dindar and Partners, Mpumalanga
  - Private Practice - Cathy Spargo, Pinelands
  - Jakaranda Hospital Pretoria, Pretoria
  - Emmed Research, Pretoria
  - Winelands Rheumatology Centre, Stellenbosch
- Spain (3):
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- United Kingdom (3):
  - Royal Sussex County Hospital, Brighton
  - Harrogate District NHS Foundation Trust, Harrogate
  - Wirral University Teaching Hospital NHS Foundation Trust, Merseyside

RESULTS

PARTICIPANT FLOW:
Groups:
- Enbrel (Etanercept): Enbrel 50mg subcutaneously every week for 24 Weeks.
  Etanercept: Head-to-head comparison
  In part 2, all subjects received 50mg subcutaneously every week from week 25-48.
- CHS-0214: CHS-0214 50mg subcutaneously every week for 24 Weeks.
  Part 2: All subjects received CHS-0214 50mg subcutaneously every week from week 25-48.
Period: Part 1
Arm/Group | Enbrel (Etanercept) | CHS-0214
Started | 323 | 324
Completed | 301 | 312
Not Completed | 22 | 12
Period: Part 2: All Subjects Receive CHS-0214
Arm/Group | Enbrel (Etanercept) | CHS-0214
Started | 280 | 284
Completed | 269 | 272
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Population: The overall number of participants is inconsistent with participant flow because of baseline characteristics analysis including both populations one and two.
Groups:
- CHS-0214: CHS-0214 50mg weekly times 24 weeks.
  CHS-0214
- Total: Total of all reporting groups
Arm/Group | Enbrel (Etanercept) | CHS-0214 | Total
Number analyzed (Participants) | 320 | 324 | 644
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 280 | 285 | 565
  >=65 years | 40 | 39 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 260 | 514
  Male | 66 | 64 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 211 | 213 | 424
  Asian | 98 | 99 | 197
  African American | 6 | 9 | 15
  Other | 5 | 3 | 8
  Not Hispanic or Latino | 307 | 313 | 620
  Hispanic or Latino | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: ACR-20 - 20% Improvement According to American College of Rheumatology Criteria
Description: The primary efficacy endpoint in Part 1 was the percentage of subjects who achieved ACR20 (20% improvement according to American College of Rheumatology criteria) at week 24 compared to baseline (last non-missing value prior to first dose). Subjects were considered an ACR20 responder if when compared to baseline (last non-missing value prior to first dose), they achieved a 20% decrease in SJC (Swollen joint count), 20% decrease in TJC (Tender joint count), and 20% improvement in 3 of the following 5 measures: high sensitivity C reactive protein(hs-CRP), Health Assessment Questionnaire Disability Index(HAQ-DI), subjects global assessment of pain(SPA, VAS), subject's global assessment of disease activity(SGA-VAS), physician's global assessment of disease activity(PGA-VAS)
Time Frame: 24-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 256 | 256
Participants | 232 | 233

2. Secondary Outcome: ACR20 - (20% Improvement According to American College of Rheumatology Criteria) at Weeks 4, 8, 12, and 18
Description: Subjects were considered an ACR20 responder if, when compared to baseline (last non-missing value prior to first dose), they achieved a 20% decrease in SJC, 20% decrease in TJC, and 20% improvement in 3 of the following 5 measures:
  * High sensitivity C-reactive protein (hs-CRP);
  * Health Assessment Questionnaire-Disability Index (HAQ-DI);
  * Subject's global assessment of pain (ie, subject's pain assessment [SPA]-visual analog scale [VAS]);
  * Subject's global assessment of disease activity (SGA-VAS); and
  * Physician's global assessment of disease activity (PGA-VAS).
  In these calculations, the percent change from baseline to endpoint was used to determine ACR20. For percentage change calculations, results were rounded to 5 decimal places prior to comparing to the threshold of 20%.For SJCs and TJCs, the assessment of efficacy was based on mean change from baseline (last non-missing value prior to first dose evaluation).
Time Frame: Weeks 4, 8, 12 and 18
Measure: Number; unit: percentage of participants
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 323 | 324
percentage of participants
  Week 4 | 48.8 | 56.6
  Week 8 | 59.4 | 71.1
  Week 12 | 73.8 | 74.6
  Week 18 | 75 | 77.3

3. Secondary Outcome: Summary of Change in Tender Joint Count (TJC) by Study Visit
Description: The average percent improvement from baseline in individual ACR response criteria: TJC (Tender joint count) the 66/68 Joint Count evaluates 68 joints for tenderness and pain with movement. The temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeal (MCP), proximal interphalangeal (PIP), distal interphalangeal (DIP), hip, knee, ankle, tarsus, metatarsophalangeal (MTP), and interphalangeal of the feet are included in this joint count. Hip joints can be evaluated for tenderness.
Time Frame: Weeks 4,8,12,18,24,28,36,48
Population: The full analysis population differs between part one (weeks 0 to 24) and part two (weeks 25 to 48) because part two does not include the full population that began the study.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 256 | 256
Joints
  TJC - Week 4 | -9.4 (9.13) | -10.3 (9.89)
  TJC - Week 8 | -11.8 (10.00) | -13.2 (11.21)
  TJC - Week 12 | -13.9 (10.21) | -14.7 (11.05)
  TJC - Week 18 | -15.4 (10.51) | -16.4 (11.91)
  TJC - Week 24 | -16.8 (11.31) | -18.0 (12.41)
  TJC - Week 28: number analyzed (Participants) | 229 | 229
  TJC - Week 28 | -0.2 (4.39) | 0.0 (4.49)
  TJC - Week 36: number analyzed (Participants) | 229 | 229
  TJC - Week 36 | -0.5 (4.89) | 0.2 (6.39)
  TJC - Week 48: number analyzed (Participants) | 229 | 229
  TJC - Week 48 | -1.0 (5.05) | -0.4 (4.96)

4. Secondary Outcome: Summary of Change in Swollen Joint Count (SJC) by Study Visit
Description: The 66/68 Joint Count evaluates 66 joints for swelling. The temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeal (MCP), proximal interphalangeal (PIP), distal interphalangeal (DIP), hip, knee, ankle, tarsus, metatarsophalangeal (MTP), and interphalangeal of the feet are included in this joint count.
Time Frame: Weeks 4,8,12,18,24,28,36,48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 256 | 256
Joints
  Week 4 | -7.1 (7.62) | -7.3 (6.98)
  Week 8 | -8.9 (7.85) | -9.5 (7.18)
  Week 12 | -10.0 (8.09) | -10.2 (7.76)
  Week 18 | -10.7 (8.50) | -11.1 (7.98)
  Week 24 | -11.9 (8.15) | -12.3 (7.78)
  Week 28: number analyzed (Participants) | 229 | 229
  Week 28 | -0.3 (2.79) | 0.1 (3.50)
  Week 36: number analyzed (Participants) | 229 | 229
  Week 36 | -0.7 (2.96) | -0.1 (3.83)
  Week 48: number analyzed (Participants) | 229 | 229
  Week 48 | -0.9 (3.47) | -0.5 (2.90)

5. Secondary Outcome: Summary of Change in Health Assessment Questionnaire - Disability Index (HAQ-DI) by Study Visit
Description: HAQ-DI - Scales for each question range from 0-3 (0=without any difficulty; 1=with some difficulty; 2=with much difficulty; 3=Unable to do). The "total" for each category is determined by the highest score (greatest difficulty) for that category. The score for the disability index is the mean of the eight category scores. If more than 2 of the categories or 25% are missing, the scale won't be scored. If fewer than 2 or the categories are missing, the sum of the categories was divided by the number of answered categories.
Time Frame: Weeks 4,8,12,18,24,28,36,48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 256 | 256
Units on a Scale
  Week 4 | -0.313 (0.414) | -0.266 (0.391)
  Week 8 | -0.377 (0.477) | -0.401 (0.473)
  Week 12 | -0.444 (0.497) | -0.466 (0.506)
  Week 18 | -0.493 (0.532) | -0.529 (0.540)
  Week 24 | -0.594 (0.609) | -0.614 (0.556)
  Week 28: number analyzed (Participants) | 229 | 229
  Week 28 | 0.01 (0.243) | 0.03 (0.233)
  Week 36: number analyzed (Participants) | 229 | 229
  Week 36 | 0.01 (0.293) | -0.01 (0.272)
  Week 48: number analyzed (Participants) | 229 | 229
  Week 48 | -0.05 (0.279) | -0.06 (0.309)

6. Secondary Outcome: Summary of Change in Subject's Pain Assessment - Visual Analog Scale (SPA-VAS) by Study Visit
Description: The score range for the SPA-VAS is 0-100 millimeters. One total score was reported for each assessment, no subscales exist. A lower score on the left side represents a better outcome (less pain) and the higher score is on the right side representing a worse outcome (more pain).
Time Frame: Weeks 4,8,12,18,24,28,36,48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 256 | 256
Units on a scale
  Week 4 | -18.5 (22.68) | -20.2 (22.60)
  Week 8 | -23.4 (25.43) | -27.1 (22.73)
  Week 12 | -27.7 (25.86) | -29.3 (23.12)
  Week 18 | -31.8 (24.89) | -33.3 (25.31)
  Week 24 | -38.2 (22.44) | -38.1 (24.01)
  Week 28: number analyzed (Participants) | 229 | 229
  Week 28 | 1.9 (14.25) | 1.0 (12.68)
  Week 36: number analyzed (Participants) | 229 | 229
  Week 36 | 1.6 (17.16) | -0.1 (15.14)
  Week 48: number analyzed (Participants) | 229 | 229
  Week 48 | -0.9 (16.89) | -1.8 (16.99)

7. Secondary Outcome: Summary of Change in Physician's Global Assessment- Visual Assessment Scale (PGA-VAS) by Study Visit
Description: The score range for PGA-VAS is 0-100 millimeters. The patient's assessment of disease activity - with the lowest score on the left side representing "none" to the highest score on the right side representing "extremely active".
Time Frame: Weeks 4,8,12,18,24,28,36,48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Enbrel (Etanercept) | CHS-0214
Number analyzed (Participants) | 256 | 256
Units on a Scale
  Week 4 | -24.1 (19.04) | -24.3 (18.23)
  Week 8 | -29.6 (19.76) | -31.7 (19.96)
  Week 12 | -33.5 (20.99) | -35.4 (19.57)
  Week 18 | -36.3 (20.69) | -38.8 (19.60)
  Week 24 | -40.5 (19.31) | -43.2 (17.73)
  Week 28: number analyzed (Participants) | 229 | 229
  Week 28 | 0.3 (11.47) | 0.7 (8.74)
  Week 36: number analyzed (Participants) | 229 | 229
  Week 36 | -1.4 (10.75) | -0.5 (11.80)
  Week 48: number analyzed (Participants) | 229 | 229
  Week 48 | -1.9 (13.28) | -0.5 (11.47)

ADVERSE EVENTS:
Time Frame: In part one, subjects were randomized to receive either Enbrel or CHS-0214 for 24 weeks. In part two, all participants receive CHS-0214 for the remainder of the study (Weeks 25-48)
Description: Adverse events were reported for CHS-0214 and Enbrel using two arms. Part 1 (Weeks 1-24) and 2 (Weeks 25-48) were combined in reporting of adverse events, given that all subjects received CHS-0214 in Part 2. Adverse events were reported for both arms with the first arm being CHS-0214 in both parts of the study and the second arm being patients who received Enbrel in Part 1 of the study and switched to CHS-0214.
Groups:
- Enbrel-CHS-0214 (Etanercept): Enbrel 50mg weekly times 24 weeks and CHS-0214 for weeks 25 to 48.
  Etanercept: Head-to-head comparison
- CHS-0214-CHS-0214: CHS-0214 50mg weekly times 48 weeks.
  CHS-0214
Arm/Group | Enbrel-CHS-0214 (Etanercept) | CHS-0214-CHS-0214
Serious Adverse Events (participants affected / at risk) | 27/320 | 20/604
Other Adverse Events (participants affected / at risk) | 245/320 | 241/604
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enbrel-CHS-0214 (Etanercept) (N=320) | CHS-0214-CHS-0214 (N=604)
Bronchitis (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pilonidal Cyst (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Angina Unstable (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Ovarian Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Neoplasma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral Nerve Injury (Injury, poisoning and procedural complications) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocardial Ischemia (Cardiac disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 | 1
Blood Creatine Phosphokinase Increase (Investigations) | 0 | 1
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Ischemic Stroke (Nervous system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Age-Related Macular Degeneration (Eye disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enbrel-CHS-0214 (Etanercept) (N=320) | CHS-0214-CHS-0214 (N=604)
Nasopharyngitis (Infections and infestations) | 39 | 46
Urinary Tract Infection (Infections and infestations) | 17 | 22
Upper Respiratory Tract Infection (Infections and infestations) | 32 | 16
Bronchitis (Infections and infestations) | 13 | 11
Sinusitis (Infections and infestations) | 10 | 9
Cystitis (Infections and infestations) | 7 | 8
Respiratory Tract Infection - Viral (Infections and infestations) | 3 | 8
Herpes Zoster (Infections and infestations) | 5 | 7
Oral Herpes (Infections and infestations) | 10 | 7
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 11 | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Nausea (Gastrointestinal disorders) | 5 | 9
Diarrhea (Gastrointestinal disorders) | 7 | 6
Alanine Aminotransferase Increased (Investigations) | 15 | 13
Aspartate Aminotransferase Increase (Investigations) | 13 | 7
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 25 | 34
injection Site Reaction (General disorders) | 44 | 9
Headache (Nervous system disorders) | 8 | 20
Rash (Skin and subcutaneous tissue disorders) | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Hypertension (Vascular disorders) | 13 | 12
Anemia (Blood and lymphatic system disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No